CLINICAL TRIAL: NCT05860426
Title: Assessment of Confidence in the Ability to Perform Movements in Patients With Low Back Pain and Its Relationship With the Characteristics and Evolution of Pain
Brief Title: Confidence in the Ability to Perform Movements in Patients With Low Back Pain
Acronym: CONFI-LBP
Status: Completed | Type: Observational
Sponsor: Universidad de León (Other)
Responsible Party: Principal Investigator, Arrate Pinto Carral, Ph. Dr. Teacher, Universidad de León
Other Study IDs: ULE-003-2021
Record Dates: First submitted 2023-04-26; First posted 2023-05-16 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Low Back Pain
Keywords: Low Back Ache; Lumbago; Self Efficacy; Kinesiophobia; Machine Learning
MeSH Terms: conditions — Low Back Pain; Kinesiophobia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goals of this observational study are:

To determine the validity and reliability of the OPTIMAL-confidence scale in people with chronic low back pain.

To assess the influence of confidence and fear of movement on the evolution of low back pain.

The main question it aims to answer is if people with chronic low back pain present different psychoemotional variables around fear of movement and decreased confidence in their ability to perform movement that may influence their low back pain.

For this purpose, a two-phase study was designed. In the first phase, the OPTIMAL-confidence scale will be validated in patients with chronic low back pain, determining its internal consistency and validity. In the second phase, a prospective study will be carried out with patients with low back pain who attend physiotherapy centres to determine how confidence and fear of movement influence the characteristics of pain and its evolution. Data will be collected at the beginning of the physiotherapy treatment, at the end of the treatment and after three months. The data will be analysed using learning machine techniques.

DETAILED DESCRIPTION:
In the first phase of the study, a sample of patients diagnosed with chronic low back pain will bwe selected, as well as a general population of convenience. The scope of the study is the health centres of the Primary Care Management of León and El Bierzo. To calculate the optimal sample size, the criteria included in the COSMIN20 guide (Consensus-based standards for the selection of health measurement instruments) were taken into account, taking as a reference the maximum quality criterion for hypotheses testing, which states that they should be equal to or greater than 100 subjects.

The second phase will consist of a prospective observational study among patients with low back pain selected by physiotherapists and interested in participating in the study. Data will be collected at three different times: at recruitment and at the end of treatment, in person, and three months after the end of treatment, by telephone.

The scope of the study will be the Primary and Specialised Health Care Departments of León and El Bierzo.

In both cases participants will sign an informed consent form and the physiotherapists who will collect the data will be trained by researchers.

Patients will complete socio-demographic and health questions as well as validated questionnaires on confidence, self-efficacy, fear of movement, risk of chronification and disability. Participants in the second phase will complete the questionnaires not only at the beginning, but two more times.

In the validation phase of optimal-confidence, the internal consistency of the scale will be analysed, as well as convergent and known-groups validity.

In the second phase, the data will be analysed using machine learning techniques. In order to find out which variables are most influential in the evolution of low back pain, different variations of the following machine learning techniques will be used: Gaussian Naive Bayes, Complement Naive Bayes, K-Nearest Neighbours (KNN and decision trees. Experiments using oversampling techniques such as RandomOver and Smote will also be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Patients with low back pain.
* Be able to read and understand Spanish.
* Acceptance and signature of the informed consent.

Exclusion Criteria:

* Tumor and/or infection related to the back.
* Cauda equina syndrome.
* Vertebral compression fracture.
* Abdominal aneurysm.
* Central nervous system disorders.
* Confirmed diagnosis of active neoplasm.
* Presence of cognitive deficits that prevented participation in the study.
* Pregnant patients in the last year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients assigned to primary and specialized care health centers in the province of Leon (Spain), who were diagnosed with low back pain by their referring physician.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Confidence at 3 months | Recruitment, "physiotherapy discharge" (week 3) and 3 months later.
  Outpatient Physical Therapy Improvement in Movement Assessment Log (OPTIMAL) instrument, confidence scale, spanish version. Total score ranges from 0-100 points, with higher scores indicating worse outcome (lower confidence).

SECONDARY OUTCOMES:
Change from Baseline Kinesiophobia at 3 months. | Recruitment, "physiotherapy discharge" (week 3) and 3 months later.
  Tampa scale of kinesiophobia (TSK-11), spanish version. Total score ranges from 11-44 points, with higher scores indicating worse outcome (greater fear).
Change from Baseline Disability at 3 months. | Recruitment, "physiotherapy discharge" (week 3) and 3 months later.
  Oswestry disability index (ODI), spanish version. Total score ranges from 0-100 points, with higher scores indicating worse outcome (greater disability).
Change from Baseline Risk at 3 months. | Recruitment, "physiotherapy discharge" (week 3) and 3 months later.
  STart Back screening tool (SBST-9), spanish version. Total score ranges from 0-9 points, with higher scores indicating worse outcome (greater risk).
Change from Baseline Intensity of pain at 3 months. | Recruitment, "physiotherapy discharge" (week 3) and 3 months later.
  Numerical Pain Rating Scale (NPRS). Total score ranges from 0-10 points, with higher scores indicating worse outcome (higher pain).

OTHER OUTCOMES:
Self-Efficacy. | Recruitment.
  Chronic Pain Self-efficacy scale, spanish version. Total score ranges from 0-100 points, with higher scores indicating better outcome (higher efficacy).
Socio-demographic information. | Recruitment.
  age, sex, area of residence, marital status, educational level, employment status, weight, height, chronic diseases, treatments, frequency of physical activity, walking assistance, location of pain, sleep disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Arrate Pinto-Carral, Ph Dr, Study Director — Universidad de León; Mª José Álvarez-Álvarez, Ph Dr, Study Director — Universidad de León
Locations (1):
- University of León, Ponferrada, León, Spain

IPD SHARING:
Plan to Share IPD: No
For safety, the researchers only plan to use the data collected as a whole and prefer to safeguard the database generated only for this research. However, it could be made available to other researchers upon request for justified purposes such as new studies.

REFERENCES:
- [Background] Delitto A, George SZ, Van Dillen L, Whitman JM, Sowa G, Shekelle P, Denninger TR, Godges JJ; Orthopaedic Section of the American Physical Therapy Association. Low back pain. J Orthop Sports Phys Ther. 2012 Apr;42(4):A1-57. doi: 10.2519/jospt.2012.42.4.A1. Epub 2012 Mar 30. PMID 22466247
- [Background] George SZ, Fritz JM, Silfies SP, Schneider MJ, Beneciuk JM, Lentz TA, Gilliam JR, Hendren S, Norman KS. Interventions for the Management of Acute and Chronic Low Back Pain: Revision 2021. J Orthop Sports Phys Ther. 2021 Nov;51(11):CPG1-CPG60. doi: 10.2519/jospt.2021.0304. PMID 34719942
- [Background] Guccione AA, Mielenz TJ, Devellis RF, Goldstein MS, Freburger JK, Pietrobon R, Miller SC, Callahan LF, Harwood K, Carey TS. Development and testing of a self-report instrument to measure actions: outpatient physical therapy improvement in movement assessment log (OPTIMAL). Phys Ther. 2005 Jun;85(6):515-30. PMID 15921473
- [Background] Pinto-Carral A, Fernandez-Villa T, Guccione AA, Cuadrado FM, Cancela JM, Molina AJ. Validity, Reliability, and Responsiveness of the Spanish Version of the OPTIMAL Instrument. PM R. 2019 Mar;11(3):258-269. doi: 10.1016/j.pmrj.2018.05.021. Epub 2019 Jan 22. PMID 29860022
- [Background] Deyo RA, Dworkin SF, Amtmann D, Andersson G, Borenstein D, Carragee E, Carrino J, Chou R, Cook K, DeLitto A, Goertz C, Khalsa P, Loeser J, Mackey S, Panagis J, Rainville J, Tosteson T, Turk D, Von Korff M, Weiner DK. Report of the NIH Task Force on research standards for chronic low back pain. Pain Med. 2014 Aug;15(8):1249-67. doi: 10.1111/pme.12538. PMID 25132307
- [Background] Gusi N, del Pozo-Cruz B, Olivares PR, Hernandez-Mocholi M, Hill JC. The Spanish version of the "STarT Back Screening Tool" (SBST) in different subgroups. Aten Primaria. 2011 Jul;43(7):356-61. doi: 10.1016/j.aprim.2010.05.019. Epub 2011 Feb 5. PMID 21296465
- [Background] Hill JC, Dunn KM, Lewis M, Mullis R, Main CJ, Foster NE, Hay EM. A primary care back pain screening tool: identifying patient subgroups for initial treatment. Arthritis Rheum. 2008 May 15;59(5):632-41. doi: 10.1002/art.23563. PMID 18438893